

# NON-INTERVENTIONAL STATISTICAL ANALYSIS PLAN FOR SECONDARY DATA COLLECTION STUDY

# Non-Interventional Study Protocol C2661041

Multinational Retrospective Chart Review Study to Assess the Characteristics, Treatment Outcomes and Resource Use among Adult Patients Hospitalised for Community-Acquired Pneumonia (CAP) and Complicated Skin or Soft Tissue Infections (cSSTI) Treated with Zinforo® (ceftaroline fosamil) in a Usual Care Setting

Statistical Analysis Plan (SAP)

**Version**: FINAL v2.0

Author: PPD

**Date**: 3- Dec-2020

# **TABLE OF CONTENTS**

| 2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>HY | STUDY DESIGN STUDY POPULATION DATA SOURCE STUDY OBJECTIVES | 6<br>8 |
|---|---|---|
| 2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>HY | STUDY DESIGN | 6<br>8 |
| 2.1.3<br>2.1.4<br>HY | STUDY POPULATION | 6<br>8 |
| 2.1.4<br><b>HY</b> | STUDY OBJECTIVES | |
| HY | | 8 |
| | POTHECES AND DECISION DIVINES | |
| | POTHESES AND DECISION RULES | 9 |
| 3.1.1 | STATISTICAL HYPOTHESES | 9 |
| 3.1.2 | | |
| AN. | ALYSIS SETS/POPULATIONS | 9 |
| 4.1.1 | FULL ANALYSIS SET | 9 |
| 4.1.2 | | |
| 4.1.3 | OTHER ANALYSIS SET | 9 |
| 4.1.4 | SUBGROUPS | 9 |
| EN | DPOINTS AND COVARIATES | 10 |
| 5.1.1 | Effectiveness outcomes | 10 |
| 5.1.2 | TREATMENT RESPONSE TO ZINFORO® | 10 |
| 5.1.3 | | |
| 5.1.4 | | |
| STA | ATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 16 |
| 7.1.1 | | |
| - | | |
| LIS | T OF TABLES AND TABLE SHELLS | 18 |
| 8.1.1 | | |
| 8.1.2 | CHARACTERISTICS OF PATIENTS WITH CAP | 18 |
| | 3.1.1 3.1.2 AN. 4.1.1 4.1.2 4.1.3 4.1.4 EN. 5.1.1 5.1.2 5.1.3 5.1.4 5.1.5 5.1.6 5.1.7 5.1.8 HA STA 7.1.1 7.1.2 7.1.3 7.1.4 7.1.5 LIS 8.1.1 | ANALYSIS SETS/POPULATIONS |

| 0 | DFI | FEDENCES | Q1 |
|---|---|---|---|
| | 8.1.14 | TREATMENT MODIFICATIONS / ADVERSE EVENTS IN PATIENTS WITH CSSTI | . 77 |
| | 8.1.13 | ADDITIONAL CLINICAL OUTCOMES IN PATIENTS WITH CSSTI | |
| | 8.1.12 | TREATMENT RESPONSE TO ZINFORO® IN PATIENTS WITH CSSTI | |
| | HOPSPI | TALIZATION IN PATIENTS WITH CSSTI | |
| | 8.1.11 | | |
| | 8.1.10 | HEALTHCARE RESOURCE USE FOR CSSTI PATIENTS STARTING ZINFORO | . 59 |
| | 8.1.9 | PATIENT CHARACTERISTICS IN PATIENTS WITH CSSTI | . 50 |
| | 8.1.8 | ANALYSES OF CSSTI PATIENTS | . 50 |
| | 8.1.7 | TREATMENT MODIFICATIONS / ADVERSE EVENTS IN PATIENTS WITH CAP | . 43 |
| | 8.1.6 | ADDITIONAL CLINICAL OUTCOMES IN PATIENTS WITH CAP | . 42 |
| | 8.1.5 | TREATMENT RESPONSE TO ZINFORO® IN PATIENTS WITH CAP | . 41 |
| | HOPSPI | TALIZATION IN PATIENTS WITH CAP | . 35 |
| | 8.1.4 | PHYSICIANS USE OF ZINFORO® (AND OTHER ANTIBIOTICS) DURING INDEX | |
| | 8.1.3 | HEALTHCARE RESOURCE USE FOR PATIENTS WITH CAP STARTING ZINFORO | . 26 |

# LIST OF TABLES

| Table 1. Demographic characteristics of included CAP patients at index hospitalization | n 18 |
|---|---|
| Table 2. Medical history in patients with CAP | . 20 |
| Table 3. Hospitalization and treatments in the 3 months prior to index hospitalization i | n |
| patients with CAP | . 21 |
| Table 4. Diagnostics in patients with CAP | . 22 |
| Table 5. Diagnosis and infection details in patients with CAP | . 23 |
| Table 6. Microbiological findings in patients with CAP | |
| Table 7. Additional tests and vaccination status in patients with CAP | . 25 |
| Table 8. Utilization during index hospitalization in patients with CAP | . 26 |
| Table 9. Hospitalisation cost in patients with CAP | |
| Table 10. Utilization during index hospitalization by response status in patients with C | AP |
| Table 11. Hospitalisation cost by response status in patients with CAP | |
| Table 12. Ventilation and parenteral nutrition in patients with CAP | |
| Table 13. Treatments received during index hospitalization in patients with CAP | |
| Table 14. Complications during index hospitalization in patients with CAP | |
| Table 15. Dosages of Zinforo and other antibiotics in patients with CAP | |
| Table 16. Resource use post index hospitalization in patients with CAP | |
| Table 17. Pre Zinforo treatment- Summary across all treatment lines in patients with C | |
| Table 18. Pre Zinforo treatment by line of treatment in patients with CAP | |
| Table 19. Zinforo treatment during index hospitalization in patients with CAP | |
| Table 20. Zinforo administered in combination therapy in patients with CAP | |
| Table 21. Zinforo treatment and concomitant therapy in patients with CAP | |
| Table 22. Response to Zinforo treatment in patients with CAP | |
| Table 23. Additional clinical outcomes in response to Zinforo treatment in patients wit | |
| CAP | |
| Table 24. Clinical failure with Zinforo in patients with CAP | |
| Table 25. Clinical failure with Zinforo due to adverse events in patients with CAP | |
| Table 26. Seriousness of adverse events in patients with CAP | |
| Table 27. Post Zinforo treatment- Summary across all lines in patients with CAP | |
| Table 28. Response to post-Zinforo treatment in patients with CAP | |
| Table 29. Demographic characteristics of included cSSTI patients at index hospitalizat | |
| Table 30. Medical history in patients with cSSTI | |
| Table 31. Hospitalization and treatments in the 3 months prior to index hospitalization | . in |
| patients with cSSTI | . 53 |
| Table 32. cSSTI Characteristics | |
| Table 34. Diagnosis and infection details in patients with cSSTI | |
| Table 35. cSSTI Diagnostics | |
| Table 37. Utilization during index hospitalization in patients with cSSTI | |
| Table 38. Hospitalisation cost in patients with cSSTI | . 60 |

Table 39. Utilization during index hospitalization by response status in patients with Table 42. Treatments received during index hospitalization in patients with cSSTI ...... 64 Table 43. Complications during index hospitalization in patients with cSSTI...... 65 Table 46. Pre Zinforo treatment- Summary across all treatment lines in patients with cSSTI 68 Table 48. Zinforo treatment during index hospitalization in patients with cSSTI......71 Table 52. Additional clinical outcomes in response to Zinforo treatment in patients with Table 54. Clinical failure with Zinforo due to adverse events in patients with cSSTI..... 78 Table 56. Post Zinforo treatment- Summary across all lines in patients with cSSTI....... 81 

# 1 AMENDMENTS FROM PREVIOUS VERSION(S)

Not applicable.

#### 2 INTRODUCTION

Community-acquired pneumonia (CAP) is a common respiratory illness, involving an acute infection of the lungs. <sup>1-6</sup> CAP is associated with considerable morbidity, mortality, <sup>5,7,8</sup> resource use and healthcare costs. <sup>2,4,8,9</sup> Complicated skin and soft-tissue infections (cSSTI) include infected ulcers, infected burns and major abscesses that require hospitalization and represents a major clinical problem <sup>10-12</sup> as they are also associated with considerable morbidity, mortality, resource use and healthcare costs. <sup>13-17</sup> Current treatment options for cSSTI are compromised by resistance in particular countries and tolerability issues. In patients with CAP or cSSTI (particularly those at risk of treatment failure), there is a need for an alternative treatment option that will improve empiric treatment success rates by providing activity against a range of suspected causative pathogens (including methicillin-resistant *S. aureus* (MRSA) and S. *pneumoniae*) combined with a good tolerability profile.

Ceftaroline fosamil (Telflaro in the United States [US]; Zinforo® ex-US) is a novel 5th generation cephalosporin with rapid bactericidal action against a broad range of common Gram positive and Gram negative pathogens. Zinforo® is approved in the European Union (EU) in adults and children from time of birth for the treatment of cSSTI and CAP. The recommended treatment duration for cSSTI is 5 to 14 days and the recommended duration of treatment for CAP is 5 to 7 days.

Zinforo® is an effective treatment for patients hospitalised with CAP or cSSTI, including those at risk of treatment failure and/or with intolerance/contraindications to commonly-used antibiotics. <sup>18-26</sup> At present, the real-world use and effectiveness of Zinforo® in treating patients hospitalized with CAP and cSTTI has not been evaluated in a usual care setting in Europe and Latin America.

#### 2.1.1 STUDY DESIGN

This is a multinational, multicentre, observational, retrospective cohort study. The hospital medical records of patients with cSSTI or CAP treated with Zinforo® in a usual care setting and who meet the eligibility criteria will be reviewed. For eligible patients, relevant data will be extracted from the hospital medical records from 3-months before the date of the index hospital admission until 30-days after the hospital discharge date or death, whichever occurs first.

#### 2.1.2 STUDY POPULATION

Patients must meet all of the following inclusion criteria to be eligible for this study:

1. Age 18 years or older at admission date to the hospital.

- 2. Received four (4) or more consecutive IV doses of Zinforo® in usual care on or before 31-May-2019.
- 3. Admitting diagnosis to the hospital was either CAP or cSSTI (see diagnostic criteria as specified in the study protocol).

Patients meeting any of the following exclusion criteria are not eligible for this study:

- 1. Patients who were participating in an interventional clinical trial during the same hospital admission in which Zinforo® was administered
- 2. Patients whose hospital medical records are missing documentation of the diagnostic criteria for either cSSTI or CAP
- 3. Patients whose hospital medical records are missing details of dosing with Zinforo®
- 4. Patients whose hospital medical records are missing information on the success/failure of Zinforo® treatment and the reason why treatment was discontinued
- 5. Patients whose hospital medical records are missing discharge date and status information.

## **CAP-specific Exclusion Criteria:**

• Patients admitted hospital for another medical condition who developed signs and symptoms of hospital-acquired pneumonia (HAP) or ventilator-associated pneumonia (VAP) 48-hours or more after the admission date are not eligible for this study.

#### cSSTI-specific Exclusion Criteria:

- Patients with uncomplicated SSTI are not eligible for this study.
- Patients with skin and soft tissue infection complicated by the presence of orthopedic or joint replacement prostheses are not eligible for this study.
- Patients with known or suspected endocarditis, osteomyelitis, or septic arthritis are not eligible for this study

Hospital sites participating in this study will identify all patients who were dispensed four or more intravenous (IV) doses of Zinforo® in usual care on or before 31-May-2019 by querying their hospital pharmacy dispensing records. Potentially eligible patients treated with Zinforo® for either CAP or cSSTI will be identified by querying hospital discharge records for diagnosis codes indicative of either CAP or cSSTI using the World Health Organization International Classification of Diseases 10th revision (ICD-10; see Annex 3 for the list of ICD-10 codes). The hospital medical records of potentially eligible patients treated with Zinforo® will be screened manually by site staff to identify the subset of eligible CAP and cSTTI patients who meet all inclusion criteria without meeting any of the exclusion criteria.

#### 2.1.3 DATA SOURCE

Data for this study are collected by a retrospective medical chart extraction from participating hospitals in Europe and Latin America that have treated patients with CAP or cSSTI in usual care during the study period. All data are entered by sites into electronic case report forms (eCRFs). De-identified data are collected following the Health Insurance Portability and Accountability Act (HIPAA)-compliant safe harbor approach.

#### 2.1.4 STUDY OBJECTIVES

The overall study aim of this study is to provide real world evidence (RWE) on the characteristics, clinical management, treatment outcomes and healthcare resource use of adult patients aged 18 years and older admitted to the hospital for CAP or cSSTI who received Zinforo® in a usual care setting in Europe and Latin America on or before 31-May-2019.

Specific objectives of this study are to analyze for the CAP and cSSTI cohorts:

- Objective 1 "Patient characteristics": To describe the characteristics of patients hospitalized for CAP or cSSTI who received Zinforo® in a usual care setting in Europe and Latin America on or before 31-May-2019
- Objective 2 "Use of Zinforo": To describe physicians' use of Zinforo® in the clinical management of patients hospitalized for CAP or cSSTI in relation to their use of other antibiotics (first-line vs. second-line/salvage, monotherapy vs. combination therapy, empiric vs. definitive therapy)
- Objective 3 "Clinical response": To estimate the proportion of patients hospitalized for CAP or cSSTI who responded to Zinforo® (clinical response defined as no further intravenous (IV) antibiotic, switch to an oral antibiotic, or IV antibiotic treatment streamlining/de-escalation prior to discharge from the hospital);
- Objectives 4 "Additional clinical outcomes": To describe the clinical outcomes (eg, hospital readmission, mortality) of patients hospitalized for CAP or cSSTI after starting Zinforo® stratified by clinical response;
- Objective 5 "Treatment modification": To estimate the proportion of patients hospitalized for CAP or cSSTI who had treatment modification of Zinforo® (defined as switch to another IV antibiotic due to an adverse reaction, drugdrug interaction, insufficient response or a microbiological diagnosis indicating that the pathogen is not susceptible to Zinforo®)
- Objective 6 "Healthcare resource use": To describe the healthcare resource use of patients hospitalized for CAP or cSSTI after starting Zinforo® stratified by clinical response.

#### 3 HYPOTHESES AND DECISION RULES

This study is purely descriptive in nature and there are no a priori hypotheses specified. Hence, no statistical tests or formal statistical inference will be performed.

# 3.1.1 STATISTICAL HYPOTHESES

Not applicable.

#### 3.1.2 STATISTICAL DECISION RULES

Not applicable.

#### 4 ANALYSIS SETS/POPULATIONS

#### 4.1.1 FULL ANALYSIS SET

The data set will be split by the type of infection (CAP, cSSTI) into two separate analyses sets. The analyses will be performed separately for each of these data sets which will include all subjects with the respective type of infection who are eligible for the study and whose data was entered into the study database (see Section 2.1.1 for eligibility criteria).

#### 4.1.2 SAFETY ANALYSIS SET

Not applicable.

#### 4.1.3 OTHER ANALYSIS SET

No other analysis data sets will be defined.

#### 4.1.4 SUBGROUPS

For selected outcomes, subgroup analyses will be conducted by geography (Europe including Russia, Latin America).

Certain outcomes will be stratified by covariates of interest provided each of the strata exceeds the minimum sample size of 30 patients (5% of total) as specified in the protocol. Covariates for stratified analyses will include:

- For cSSTI patients: Early response within 3 days
- For CAP patients: Early response within 4 days
- Line of treatment
- Age: >65 or  $\le 65$

#### 5 ENDPOINTS AND COVARIATES

#### 5.1.1 EFFECTIVENESS OUTCOMES

### 5.1.2 TREATMENT RESPONSE TO ZINFORO®

As described in the protocol the clinical response is measured according to the following widely accepted criteria:

- CAP patients: demonstrating clinical stability (defined according to the IDSA guidelines as temperature of ≤37.8 °C, heart rate of ≤100 beats/min, respiratory rate of ≤24 breaths/min, systolic blood pressure of ≥90mmHg, oxygen saturation of ≥90%, and confusion/disorientation recorded as absent) and clinical improvement (defined as improvement of at least 1 of 4 symptoms present at baseline (i.e., cough, dyspnea, pleuritic chest pain, sputum production) with worsening of none.)
- cSSTI patients: ≥20% reduction from baseline infection area and cessation of spread measured by total infection area

Making referencing to the definitions above the following variables will be extracted from charts to assess the clinical response to Zinforo® treatment received during index hospitalization:

- Clinical response, Yes / No, dichotomous from CRF
  - o If "Yes", time to clinical response
- Clinical Cure, Yes / No, dichotomous from CRF
  - o If "Yes", time to clinical cure
- Clinical failure defined as any one of the following:
  - Treatment modification due to adverse event (AE)
  - Time to modification (days from treatment initiation)
  - o Drug-drug interaction
  - o Insufficient response (followed by switch)
  - O Death due to index infection
  - o Death due to other cause
  - o Relapse or recurrence

For CAP patients specifically, the following effectiveness outcomes will be assessed:

- Time to clinical stability (according to the guidelines from the Infectious Disease Society of America, (IDSA))
- Time to clinical improvement (defined as improvement of at least 1 of 4 symptoms present at baseline)

For cSSTI patients specifically, the following effectiveness outcomes will be assessed:

• Time to >20% reduction from baseline infection area


CCI

- - Time to cessation of spread measured by total infection area
  - Time to cessation of spread measured by infection length and width
    - o oral switch,
    - o time to symptom resolution,
    - o time to clinical stability (Halm criteria),
    - o time to oral switch.

The following effectiveness endpoint on early response will be calculated based on the abstracted information:

### For cSSTI patients:

- Time to clinical response: Calculated as maximum of:
  - o Time to ≥20% reduction from baseline infection area
  - o Time to cessation of spread measured by total infection area
  - o Time to cessation of spread measured by infection length and width
- Early response within 3 days (3 levels):
  - 1: Response according to dichotomous CRF item = "Yes" AND time to response ≤ 3 days
  - o 2: Response = "Yes" AND time to response >3 days
  - o 3: No response according to dichotomous CRF item

### For CAP patients:

- Time to clinical response: Calculated as maximum of:
  - o Time to clinical stability
  - o Time to clinical improvement
- Early response within 4 days (3 levels):
  - 1: Response according to dichotomous CRF item = "Yes" AND time to response ≤ 4 days
  - o 2: Response = "Yes" AND "Time to response" > 4 days
  - o 3: No response according to dichotomous CRF item

### 5.1.3 ADDITIONAL CLINICAL OUTCOMES

- Discharge status
- Rehospitalization within 30 days after discharge
- Vital status 30 days after discharge

#### Etiology of clinical failure is also assessed:

- Minimum inhibitory concentrations (MIC) of antibacterial drugs
  - o Day of assessment since index hospitalization
  - o MIC of ceftaroline for all isolated pathogens

- o MIC of oxacillin, vancomycin, linezolid, and daptomycin for S. aureus
- o MIC of ceftriaxone for MSSA
- o MIC of penicillin and ceftriaxone for S. pneumonia

#### 5.1.4 TREATMENT MODIFICATIONS / AE

The following variables are extracted from charts of eligible patients to assess proportion of patients who had treatment modification of Zinforo® treatment:

- Treatment switch to another IV antibiotic due to adverse event (AE)
- Drug-drug interaction
- Insufficient response
- Microbiological diagnosis

AEs resulting in treatment modification are also collected:

- o Infections and infestations
- o Blood and lymphatic system disorders
- o Immune system disorders
- o Nervous system disorders
- Vascular disorders
- Gastrointestinal disorders
- Hepatobiliary disorders
- o Renal urinary disorders
- o General disorders and administrative site conditions
- Investigations
- o Other
- Seriousness of AE
- Type of criteria applied to assess seriousness of AE

#### 5.1.5 OTHER ENDPOINTS

Beyond the range of effectiveness endpoints specified above (sections 5.1.1), the additional outcomes listed below will be analysed.

#### 5.1.6 PATIENT CHARACERISTICS AT INDEX HOSPITALIZATION

The following variables on patient characteristics are collected from the patient charts:

- Patient demographics at index hospitalization
  - Year of patient hospitalization
  - o Sex
  - o Age category: >65 and ≤65 years
  - Country
  - o Race, ethnicity


انانا

- - o Height (cm)
  - Weight (kg)
  - o Patient's type of residence/cohabitation
  - Smoking habits
  - Medical history of patients treated with Zinforo®
    - Medical conditions that the patient presented with at index visit hospitalization
    - O Hospitalization for any reason in the 3 months before the index visit
    - Invasive major surgical treatment in the 3 months before the index visit hospitalization
    - Therapies in the 3 months before the index visit hospitalization
      - Antimicrobial (e.g. antibiotics, antivirals)
      - Immunosuppressors/ immunomodulators
      - Anticoagulants
      - Non-steroid anti-inflammatory agents (NSAIs)
      - Home infusion therapy
      - Home wound care provided by a medical professional
  - CAP-specific characteristics
    - o Radiographic findings
    - o Triggering signs and symptoms at diagnosis
    - o Severity of CAP
    - o Prognostic Scoring system
    - Time of CAP diagnosis
    - o Recurrence of infection
    - o Microbiologic diagnosis / type of investigation performed
    - o PCF determination of H1N1 influence virus
    - o Influenca vaccination status (12 month pre index)
    - o Pneumococcal vaccination status
    - o Biomarkers used for monitoring
  - cSSTI-specific characteristics
    - o Type of lesion involved
    - o Type of body area involved
    - o Extension of the skin infection in (sqcm)
    - o Level of infection
    - o Anatomical structures that were affected
    - o Time of c SSTI diagnose
    - o Recurrence of infection?
    - o Triggering signs and symptoms at diagnosis
    - o Systemic signs of cSSTI diagnosis
    - o Diagnostic tests performed

- Microbiological diagnosis
- o Methicillin susceptible S. aureus (MSSA)

# 5.1.7 PHYSICIANS' USE OF ZINFORO® DURING INDEX HOSPITALIZATION

- Pre Zinforo® treatment
  - Antibiotic class
  - Line of therapy
  - o Route of administration
  - o Duration of treatment Time from admission to 1st dose
  - Time from symptom onset to 1st dose
  - Treatment type
  - o Daily dose
  - o Treatment modified (Reason)
  - o Treatment response/ failure
  - o Time to clinical response / failure
  - o Clinical failure details
- Zinforo® treatment
  - Duration of treatment
  - o Time from admission to 1st dose
  - o Time from symptom onset to 1st dose
  - Treatment type
  - o Daily dose
  - o Number of infusions per day
  - o Administration location
  - Zinforo® as monotherapy/ combination (including further details of combination therapy)
  - Concomitant therapy
- Post Zinforo® antibiotic treatment
  - o Generic name of treatment
  - o Line of therapy
  - o Route of administration
  - o Time from Zinforo® discontinuation to initiation of new treatment
  - o Daily dose
  - Number of doses administered
  - o Administration location
  - o Reason for switch to this treatment:
  - Treatment response
  - o Clinical cure achieved?
  - o Clinical failure details

# 5.1.8 HEALTHCARE RESOURCE USE AND COST FOR PATIENTS STARTING ZINFORO®

The following variables are collected in the CRF on the resource utilization for patients starting Zinforo® during index hospitalization:

- Duration of index hospitalization
- Duration in intensive care unit during index hospitalization
- Renal replacement therapy initiated after initiating Zinforo®
- Treatments (Surgery / blood pressure support) during index hospitalization
- Home-based care through a health-care agency (e.g. for wounds, intravenous infusions), nursing services, etc. after discharge (days)
- Re-hospitalization within 30 days of initial discharge:
  - o Number of times and days
  - o Reason: Index infection, other
- Development of sepsis during index hospitalization
  - o Sepsis
    - Severe sepsis
    - Septic shock
- Patient treatment during index hospitalization
  - Quick sepsis-related organ failure assessment (qSOFA) conducted at the time of the index hospitalization admission:
  - o Patient requiring isolation
  - o Patient requiring mechanical ventilation
  - o Patient requiring oxygen therapy
  - o Patient requiring parenteral nutrition
  - O Patient suffer acute renal failure necessitating renal replacement therapy during index
  - Patient receiving during index therapy surgery or blood pressure support
- Total doses of Zinforo®
- Total dose of other antibiotics in combination therapy with Zinforo®
- Total doses of other antibiotics post Zinforo® treatment

To get an indication for the economic impact related to the treatment of CAP and cSSTI approximate hospitalization cost will be calculated based on the calculated sum of hospital days and a list of country specific per diem rates. To assess a range of the cost and depending on the data available from each of the countries two per diem rates will be used for the cost calculation: The average per diem rate of hospitals providing standard services for these type of infections and average per diem rate of hospitals providing the highest level of medical services. "Standard" or secondary level hospitals are anticipated to be institutions that are primarily treating referral cases, with bed size ranging from 200

to 800 beds. Advanced or tertiary-level/teaching hospitals will be typically comprise hospitals intended for referral cases, with a teaching component and highly specialised staff and technical equipment, including ICU and bed size ranging from 300 to 1,500 beds. The cost estimates will be expressed in both national currency as well as in USD using sector specific exchange rate or power purchasing parities:

- Country specific calculation of approximate hospitalization cost:
  - Cost assuming a standard level hospital
     Total hospital cost= total number of bed days \* per diem rate standard hospital (local currency / USD)
  - Cost of advanced level hospitals
     Total hospital cost= total number of bed days \* per diem rate advanced hospital (local currency / USD)

#### 6 HANDLING OF MISSING VALUES

No imputation for missing values will be performed. Missing values will be tabulated in the descriptive tables.

#### 7 STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

#### 7.1.1 SAMPLE SIZE

Given that this study is purely descriptive in nature and since there are no a priori hypotheses specified, a formal sample size calculation is not applicable. It is anticipated that approximately 600 eligible CAP and cSSTI patients from 35-40 participating sites will be sufficient to conduct this study.

#### 7.1.2 STATISTICAL METHODS

All study outcomes (effectiveness, clinical outcomes, and other endpoints) will be analysed using descriptive statistics to summarize patient and disease characteristics, treatment patterns, and treatment outcomes and health care resource utilisation. Means, standard deviations, medians, minimums and maximums will be provided for continuous variables when performing descriptive analysis of continuous data. Absolute counts and percentages will be provided when performing descriptive analysis of categorical data.

The following variables will be calculated from the information collected in the CRF:

- Body mass index (BMI): Weight(kg) / (Height(cm)\*0.01)<sup>2</sup>
- Geographic region, 2 levels:
  - o 1: Europe (France, Greece, Italy, Spain, Russia)
  - o 2: Latin America (Brazil, Columbia, Mexico)

Data analyses will be performed separately for the two patient cohorts: CAP and cSSTI. No analyses combining these two patient cohorts will be performed.

Within these patient groups data will be presented in aggregate, as well as stratified by patient and disease characteristics of interest, such as geographic region (see section 4.1.4).

Due to the descriptive nature of the analyses no formal statistical tests will be conducted.. All statistical analyses will be executed using statistical software SAS version 9.4 or later.

# 7.1.3 STATISTICAL ANALYSES

## 7.1.4 SPECIFIC APPROACH

Using the endpoints described in section 5.1.6, patient characteristics will be described by summarizing patient demographics at index hospitalization, as well as patient's medical history. CAP-specific characteristics and cSSTI-specific characteristics will also be summarized for each patient cohort respectively. To describe physicians' use of Zinforo® in the clinical management of the patients hospitalized for CAP or cSSTI, details on pre-Zinforo treatment, Zinforo treatment as well as post-Zinforo antibiotic treatment will be summarized to describe line of therapy, monotherapy vs. combination therapy, etc (see related endpoints described in section 5.1.7). Proportion of patients with a clinical response, clinical cure and clinical failure in response to Zinforo® treatment will be summarized. Using the endpoints outlined in section 5.1.3, the clinical outcomes (e.g. hospital readmission, mortality) of patients hospitalized for CAP or cSSTI after starting Zinforo will be summarized and stratified by clinical response. Treatment modification Zinforo® and reasons for treatment modification will be described for the CAP and cSSTI patient cohorts, using the endpoints collected as described in section 5.1.4. Healthcare resource utilization will be described for patients hospitalized for CAP or cSSTI after starting Zinforo® and stratified by clinical response, using the appropriate endpoints as described in section 5.1.8.

#### 7.1.5 INTERIM ANALYSIS

One interim analysis will be performed on all validated and locked patient data within the EDC. The time frame for the interim database lock and interim analysis will be based on Pfizer's internal needs and dissemination plans. The interim analysis will be performed on the full set of planned analyses. Due to the purely descriptive nature of the study no further considerations on issues such as alpha spending are required. The final analyses will be performed after completion of data collection and subsequent data base lock.

### 8 LIST OF TABLES AND TABLE SHELLS

### 8.1.1 ANALYSES OF PATIENTS WITH CAP

## 8.1.2 CHARACTERISTICS OF PATIENTS WITH CAP

# Table 1. Demographic characteristics of included CAP patients at index hospitalization

| CAP Demographic characteristics | All CAP patients (N=XX) |
|---------------------------------|-------------------------|
| | n % |

#### Age

<90 years

≥ 90 years

If <90 years, Mean (SD)

Median (Min Max)

<65 years

≥ 65 years

#### Sex

Male

Female

#### Race, Ethnicity

White, Caucasian

Black/African-American/Caribbean

Latin-American

Asian

Middle Eastern

Mixed

Other

Not available

## Country

France

Greece

Italy

Spain

Russia

Brazil

Columbia

Mexico

### **CAP Demographic characteristics**

All CAP patients (N=XX)
n %

#### Height (cm)

Mean (SD)

Median (Min-Max)

Unknown

### Weight (kg)

Mean (SD)

Median (Min-Max)

Unknown

#### BMI

Mean (SD)

Median (Min-Max)

Unknown

# Type of residence/cohabitation (pre index

if changed after discharge)

Nursing home or extended care facility

Living independently

Living with care support (family, friend, hired support)

Other

Unknown

### **Smoking habits**

Non-smoker

Ex-smoker (stopped ≥ 365 days ago)

Occasional smoker (less than 1 tobacco product per day)

Habitual smoker (1 or more tobacco products per day)

Unknown

Abbreviations: n=number; SD = Standard deviation

# Table 2. Medical history in patients with CAP

| Medical history | All CAP patients (N=XX) |
|-----------------|-------------------------|
| | n % |

### Medical condition(s) at index hospitalization

None

AIDS/HIV infection

If HIV infected: Controlled with HAART

Yes (n, % of HIV infected) No (n, % of HIV infected)

Unknown (n, % of HIV infected)

Alcohol abuse

Cancer/malignancy

Cerebrovascular disease

Chronic dialysis within the past 30 days

Chronic obstructive pulmonary disease

Chronic renal disease

Congestive heart failure

Decompensated cirrhosis

Diabetes mellitus

Immunosuppressive disease

Influenza

Injection drug use

End stage liver disease

Peripheral vascular disease

Respiratory disease

Other relevant condition(s) or disease(s) requiring chronic drug

treatment.

Unknown

Abbreviations: AIDS/ HIV: acquired immunodeficiency syndrome/ human immunodeficiency virus, HAART: highly active antiretroviral therapy

# Table 3. Hospitalization and treatments in the 3 months prior to index hospitalization in patients with CAP

Prior hospitalization

All CAP patients (N=XX)

n %

# Hospitalization for any reason in the 3 months before index hospitalization

Yes

No

Unknown

If hospitalized

Duration of hospitalization previous to index

Mean (SD)

Median (Min-Max)

### Invasive major surgical treatment in the 3 months before index

Yes

No

Unknown

### Therapies received in the 3 months before index

Antimicrobial (e.g. antibiotics, antivirals)

Immunosuppressors/ immunomodulators

Anticoagulants

Non-steroid anti-inflammatory agents (NSAIs)

Home infusion therapy

Home wound care provided by a medical professional

None

# Table 4. Diagnostics in patients with CAP

CAP Diagnostic

All CAP patients (N=XX)

n %

#### Radiographic findings in tests for CAP

Infiltrate

Consolidation

Pleural effusion

Other findings

Unknown

None of the above

### Triggering signs and symptoms at CAP diagnosis

New or increased cough

Purulent sputum or change in sputum character

Auscultatory findings consistent with pneumonia

Dyspnea, tachypnea, or hypoxemia (O2 saturation < 90% on room

air or pO2 < 60 mmHg)

Fever (>38 °C oral; > 38.5 °C rectally or tympanically) or

hypothermia (< 35 °C)

WBC count > 10,000 cells/mm³ or < 4,500 cells/mm³

Unknown

None of the above

#### Criteria for severe CAP

Yes

No

Unknown

#### Prognostic scoring system used

PORT Score / Pneumonia Severity Index

Mean (SD)

Median (Min-Max)

CURB-65

Mean (SD)

Median (Min-Max)

Other

None

Unknown

Abbreviations: Max: maximum; Min: minimum; SD: standard deviation. O2: oxygen, pO2: oxygen partial pressure, WBC: white blood cells, PORT: Pneumonia Severity Index, CURB-65: Confusion, Blood urea, Respiratory rate, Blood pressure, age ≥65

# Table 5. Diagnosis and infection details in patients with CAP

| CAP Time of infection | All CAP patients (N=XX) |
|-----------------------|-------------------------|
| | n % |

# Time of CAP diagnosis

Prior to index hospitalization
Days prior to index hospitalization
Mean (SD)
Median (Min-Max)
During index hospitalization
Unknown

### **Recurrent CAP infection**

Yes No

Unknown

## Table 6. Microbiological findings in patients with CAP

**CAP Microbiological findings** 

All CAP patients (N=XX)

n %

#### Microbiological CAP diagnosis positive for

Streptococcus pneumonia

Multidrug resistant S. pneumoniae

Penicillin resistant S. pneumoniae

Escherichia coli

Mycoplasma pneumonia

Chlamydophila pneumonia

Haemophilus influenza

H. Parainfluenzae

Legionella spp.

Staphylococcus aureus

Methicillin resistance Staphylococcus aureus

Methicillin susceptible S. aureus

Gram-negative bacilli

Moraxella catarrhalis

Coxiella burnetii

Kiebsiella pneumonia

Other enterobacteria

Pseudomonas aeruginosa

Aspirative pneumonia

Other microorganism

Unknown

None of the above

### Investigation conducted for positive microbiological CAP diagnosis

Sputum examination

Blood culture

Bronchoalveolar lavage or bronchial brush examination

Pleural fluid sample examination

Legionella antigen test in urine

Pneumococcal antigen test in urine

Other

Unknown

None of the above

# Table 7. Additional tests and vaccination status in patients with CAP

| CAP test and vaccination | All CAP patients (N=XX) |
|--------------------------|-------------------------|
| | n % |

### PCF determination of H1N1 influence virus performed

Yes

No

Unknown

If yes:

Positive

Negative

# Influenza vaccination received within the 12 months pre index hospitalization

Yes

No

Unknown

#### Pneumococcal vaccination received

Yes

No

Unknown

### Biomarkers used to monitor the clinical evolution of the patient

CRP

Procalcitonin

Other biomarker

Unknown

None of the above

Abbreviation: CRP: c-reactive protein

# 8.1.3 HEALTHCARE RESOURCE USE FOR PATIENTS WITH CAP

# Table 8. Utilization during index hospitalization in patients with CAP

| | <br> | | |
|----------------------|------|----------------------|-----|
| Resource utilization | | All CAP patients (N= | XX) |
| | | n % | |

#### **Duration of index hospitalization** (days)

**STARTING ZINFORO** 

Mean (SD)

Median (Min-Max)

### **Duration of days in ICU**

Mean (SD)

Median (Min-Max)

## Quick sepsis-related organ failure assessment (qSOFA) conducted

Yes

No

Unknown

If qSOFA was conducted

(n, % of qSOFA assessed)

Glasgow coma scale <15

Systolic blood pressure <100 mmHg

High respiration rate (≥ 22 breaths per minute)

### Patient required isolation

Yes

No

Unknown

If patient isolated:

Duration of isolation (days)

Mean (SD)

Median (Min-Max)

Unknown

Abbreviations: ICU: intensive care unit; Max: maximum; Min: minimum; qSOFA: Quick sepsis-related organ failure assessment; SD: standard deviation.

# Table 9. Hospitalisation cost in patients with CAP

| Hospital Cost | All CAP patients (N=XX) |
|---------------|-------------------------|
| | n % |

# Hospital Cost - standard hospital (local currency)

Mean (SD)

Median (Min-Max)

### Hospital Cost - advanced level (local currency)

Mean (SD)

Median (Min-Max)

# Hospital Cost - standard hospital (USD)

Mean (SD)

Median (Min-Max)

# Hospital Cost - advanced level (USD)

Mean (SD)

Median (Min-Max)

Abbreviations: USD: US Dollars, Max: maximum; Min: minimum; SD: standard deviation.

# Table 10. Utilization during index hospitalization by response status in patients with CAP

| Resource utilization | CAP res<br>(N= | • | res | CAP non-<br>responders<br>(N=XX) |
|---|---|---|---|---|
| | n | % | n | % |

## **Duration of index hospitalization** (days)

Mean (SD)

Median (Min-Max)

## **Duration of days in ICU**

Mean (SD)

Median (Min-Max)

# Quick sepsis-related organ failure assessment (qSOFA) conducted

Yes

No

Unknown

If qSOFA was conducted

(n, % of qSOFA assessed)

Glasgow coma scale <15

Systolic blood pressure <100 mmHg

High respiration rate (≥ 22 breaths per

minute)

### Patient required isolation

Yes

No

Unknown

If patient isolated:

Duration of isolation (days)

Mean (SD)

Median (Min-Max)

Unknown

# Table 11. Hospitalisation cost by response status in patients with CAP

| Hospital Cost | CAP responders<br>(N=XX) | CAP non-<br>responders<br>(N=XX) |
|---------------|--------------------------|----------------------------------|
| | n % | n % |

## Hospital Cost- standard hospital (local currency)

Mean (SD)

Median (Min-Max)

# Hospital Cost- advanced level (local currency)

Mean (SD)

Median (Min-Max)

## Hospital Cost- standard hospital (USD)

Mean (SD)

Median (Min-Max)

# Hospital Cost- advanced level (USD)

Mean (SD)

Median (Min-Max)

Abbreviations: USD: US Dollars, Max: maximum; Min: minimum; SD: standard deviation.

# Table 12. Ventilation and parenteral nutrition in patients with CAP

Ventilation and parenteral nutrition

All CAP patients (N=XX)

n %

#### Patient required mechanical ventilation

Yes

No

Unknown

If patient received ventilation:

### Type of ventilation

Invasive ventilation (n, % ventilated)

Duration of invasive ventilation (days)

Mean (SD)

Median (Min-Max)

Non-invasive ventilation (n, % ventilated)

Duration of non-invasive ventilation (days)

Mean (SD)

Median (Min-Max)

Including high flow oxygen therapy

Yes (n, % ventilated)

No (n, % ventilated)

Unknown (n, % ventilated)

#### Patient received parenteral nutrition

Yes

No

Unknown

If Yes:

Duration of parenteral nutrition (days)

Mean (SD)

Median (Min-Max)

Unknown

# Table 13. Treatments received during index hospitalization in patients with CAP

Treatments received All CAP patients (N=XX) n %

### Treatment received during index hospitalization?

Surgery related to the infection

Surgery unrelated to the infection

Blood pressure support

If blood pressure support received:

Fluid resuscitation (n,% blood pressure support)

Vasopressors (n,% blood pressure support)

Invasive procedures (n,% blood pressure support)

Unknown

Other

None of the above

# Table 14. Complications during index hospitalization in patients with CAP

Complications

All CAP patients (N=XX)

n %

#### Renal failure necessitating renal replacement

Yes

No

Unknown

If renal replacement:

Duration of therapy (days)

Mean (SD)

Median (Min-Max)

Renal replacement after first dose of Zinforo

Yes (n,% with renal replacement)

No (n,% with renal replacement)

Unknown (n,% with renal replacement)

Serum creatinine at the first Zinforo dose (mg/dL)

Mean (SD)

Median (Min-Max)

Unknown

### Complications developed during index hospitalization

Sepsis

Severe sepsis

Septic shock

Unknown

None of the above

# Table 15. Dosages of Zinforo and other antibiotics in patients with CAP

Complications

All CAP patients (N=XX)

n %

#### Total number of doses of Zinforo administered

Mean (SD) Median (Min-Max)

# Total number doses of other antibiotics administered in combination with Zinforo

Mean (SD) Median (Min-Max)

# Total number of doses of other antibiotics administered post

Zinforo treatment

Mean (SD) Median (Min-Max)

# Table 16. Resource use post index hospitalization in patients with CAP

Resource utilization post index All CAP patients (N=XX) n % Home-based care received through a health-care agency (e.g. for wounds, intravenous infusions) Yes No Unknown If home based care received, Duration of home-based care (days) Mean (SD) Median (Min-Max) Re-hospitalized within 30 days of initial discharge Yes No Unknown If re-hospitalized, Number of re-hospitalizations Mean (SD) Median (Min-Max) Duration of all hospitalizations Mean (SD) Median (Min-Max) Admission reason: For index infection (n,% of re-hospitalizations) For other reason (n,% of re-hospitalizations) Unknown (n,% of re-hospitalizations)

# 8.1.4 PHYSICIANS USE OF ZINFORO® (AND OTHER ANTIBIOTICS)

DURING INDEX HOPSPITALIZATION IN PATIENTS WITH CAP

# Table 17. Pre Zinforo treatment- Summary across all treatment lines in patients with CAP

| Antibiotic treatment pre Zinforo | All CAP patients (N=XX) |
|----------------------------------|-------------------------|
| | n % |

# Antibiotic treatment for the index infection received prior to

Zinforo

Yes

No

#### Pre Zinforo treatment received

Aminoglycoside

Betalactam

Carbapenem

Ceftriaxone

Cephalosporins

Glycopeptide

Macrolide

Betalactam

/Combination

Quinolone

Sulfonamide

Clindamycin

Linezolid

Other antibiotic agent

Unknown

### Line of therapy

First

Second

Third

Fourth

### Number of pre Zinforo lines of therapy

Mean (SD)

Median (Min-Max)

# Route of administration

Oral

Intra-venous

Intra-muscular

Subcutaneous

Unknown

# **Antibiotic treatment pre Zinforo**

All CAP patients (N=XX)

n %

### **Duration of pre Zinforo treatment (days)**

Mean (SD)

Median (Min-Max)

#### Treatment type

Empiric

Definitive/Specific

Unknown

#### Number of administrations

Mean (SD)

Median (Min-Max)

### Number of doses administered

Mean (SD)

Median (Min-Max)

#### **Administration location**

ICU

General ward

At home

Out patient

Medical setting

Unknown

### **Treatment modification**

Yes

No

Unknown

If yes:

Time to treatment modification from initial dose

Reason for treatment modification

Treatment response

Time to clinical response

Clinical failure details

Daily dose unit
Table 18. Pre Zinforo treatment by line of treatment in patients with CAP

| Pre Zinforo treatment | | Line of treat | tment | |
|------------------------|----------|---------------|----------|----------|
| | 1st Line | 2nd Line | 3rd Line | 4th Line |
| | N, % | N, % | N, % | N, % |
| Aminoglycoside | | | | |
| Betalactam | | | | |
| Carbapenem | | | | |
| Ceftriaxone | | | | |
| Cephalosporins | | | | |
| Glycopeptide | | | | |
| Macrolide | | | | |
| Betalactam | | | | |
| /Combination | | | | |
| Quinolone | | | | |
| Sulfonamide | | | | |
| Clindamycin | | | | |
| Linezolid | | | | |
| Other antibiotic agent | | | | |
| Unknown | | | | |

### Table 19. Zinforo treatment during index hospitalization in patients with CAP

Zinforo treatment All CAP patients (N=XX) n %

### Zinforo line of therapy

First

Second

Third

Fourth

### **Duration of Zinforo treatment (days)**

Mean (SD)

Median (Min-Max)

Unknown

### Time from admission to 1st dose (days)

Mean (SD)

Median (Min-Max)

Unknown

### Time from symptom onset to 1st dose (days)

Mean (SD)

Median (Min-Max)

Unknown

### Treatment type

Empiric

Definitive/Specific

Unknown

### Daily dose (mg/kg)

Mean (SD)

Median (Min-Max)

### Number of infusions per day

Mean (SD)

Median (Min-Max)

Unknown

### **Administration location**

ICU

General ward

At home

Out-patient setting

Medical clinic

Unknown

Abbreviations: ICU: intensive care unit; Max: maximum; Min: minimum; SD: standard deviation.


CCI

### Table 20. Zinforo administered in combination therapy in patients with CAP

Antibiotic treatments given in combination with Zinforo

All CAP patients (N=XX)

n %

#### Zinforo as Mono/ Combination treatment

Monotherapy

Combination therapy

Unknown

If administered in combination:

### Antibiotic treatment received

Aminoglycoside

Betalactam

Carbapenem

Ceftriaxone

Cephalosporins

Glycopeptide

Macrolide

Betalactam

/Combination

Quinolone

Sulfonamide

Clindamycin

Linezolid

Other antibiotic agent

Unknown

#### Route of administration

Oral

Intra-venous

Intra-muscular

Subcutaneous

Unknown

### **Duration of combination treatment (days)**

Mean (SD)

Median (Min-Max)

Unknown

### Number of doses administered

Mean (SD)

Median (Min-Max)

Unknown

Abbreviations: Max: maximum; Min: minimum; SD: standard deviation.


# Table 21. Zinforo treatment and concomitant therapy in patients with CAP

Therapies concomitant to Zinforo

All CAP patients (N=XX)

n %

### Concomitant therapy given

Yes

No

If concomitant therapy "yes"

### Therapy received

Immunosuppressors/ Immunomodulators

Anticoagulants

Non-steroidal anti-inflammatory agents (NSAIs)

Chemotherapeutic agents

Other

Unknown

### 8.1.5 TREATMENT RESPONSE TO ZINFORO® IN PATIENTS WITH CAP

### Table 22. Response to Zinforo treatment in patients with CAP

| Treatment response | All CAP patients (N=XX) |
|--------------------|-------------------------|
| | n % |

### Zinforo treatment response

Clinical response

Clinical failure

Time to clinical response

Mean (SD)

Median (Min-Max)

Unknown

### Zinforo early treatment response

Response ≤4 days

Response >4 days

No response

Unknown

### Clinical cure achieved

Yes

No

Time to clinical cure

Mean (SD)

Median (Min-Max)

Unknown

### Clinical stability achieved

Time to clinical stability

Mean (SD)

Median (Min-Max)

Unknown

### Clinical improvement achieved

Time to clinical improvement

Mean (SD)

Median (Min-Max)

Unknown

8.1.6 ADDITIONAL CLINICAL OUTCOMES IN PATIENTS WITH CAP

# Table 23. Additional clinical outcomes in response to Zinforo treatment in patients with CAP

| With Citi | |
|------------------------------|-------------------------|
| Additional clinical outcomes | All CAP patients (N=XX) |
| | n % |

### Discharge status

Died in the hospital

Discharged to a nursing home or extended care facility

Discharged to independent living (with or without support)

Other

Unknown

### Vital status at end of follow up

Patient is still alive

Patient is deceased

If deceased

Duration of days from discharge until death(days)

Mean (SD)

Median (Min-Max)

Unknown

# Minimum inhibitory concentrations (MIC) of antibacterial drugs assessed

Yes

No

Unknown

If assessed

Day of assessment since index hospitalization

Mean (SD)

Median (Min-Max)

MIC of ceftaroline for all isolated pathogens

MIC of oxacillin, vancomycin, linezolid, and daptomycin for S. aureus

MIC of ceftriaxone for MSSA

MIC of penicillin and ceftriaxone for S. pneumonia

Abbreviations: Max: maximum; MIC: minimum inhibitory concentrations; Min: minimum; SD: standard deviation.

# 8.1.7 TREATMENT MODIFICATIONS / ADVERSE EVENTS IN PATIENTS WITH CAP

### Table 24. Clinical failure with Zinforo in patients with CAP

| Clinical failure with Zinforo | All CAP patients (N=XX) |
|-------------------------------|-------------------------|
| | n % |

### Etiology of clinical failure

Failure related to CAP Failure unrelated to CAP Unknown

#### Reason for clinical failure

Treatment modification due to AE
Time to modification (days)
Mean (SD)

Median (Min-Max)

Unknown

Drug-drug interaction

Insufficient response

Death due to index infection

Time to death due to infection (days)

Mean (SD)

Median (Min-Max)

Death due to other

Relapse or recurrence

Time to relapse/recurrence:

Mean (SD)

Median (Min-Max)

Unknown

Abbreviations: AE: adverse events; Max: maximum; Min: minimum; SD: standard deviation.

### Table 25. Clinical failure with Zinforo due to adverse events in patients with CAP

Clinical failure to Zinforo due to AEs

All CAP patients (N=XX)

n %

### AE causing Zinforo discontinuation

Infections and infestations

Clostridium difficile colitis

Other

Blood and lymphatic system disorders

Activated partial thromboplastin time (aPTT) prolonged

Agranulocytosis

Anaemia

Eosinophilia

International normalized ratio (INR) increased

Leucopenia

Neutropenia

Prothrombin time (PT) prolonged

Thrombocytopenia

Other

Immune system disorders

Anaphylaxis

Hypersensitivity (e.g. urticarial, lip and face swelling)

Pruritus

Rash

Other

Nervous system disorders

Dizziness

Headache

Other

Vascular disorders

Phlebitis

Other

Gastrointestinal disorders

Abdominal pain

Diarrhea

Nausea

Vomiting

Other

Hepatobiliary disorders

Increased transaminases

Other

Renal urinary disorders

Blood creatinine increased

Other

General disorders and administrative site conditions

Infusion site reaction (e.g. erythema, phlebitis, pain)

Pyrexia

Other

Investigations


CCI

| Clinical failure to Zinforo due to AEs | All CAP patients (N=XX) n % |
|---|---|
| Coombs direct test positive | |
| Other | |
| Unknown | |
| Abbreviations: AE: adverse events, aPTT: activated partial th | romboplastin time |

# Table 26. Seriousness of adverse events in patients with CAP

| Clinical failure to Zinforo | All CAP patients (N=XX) |
|-----------------------------|-------------------------|
| | n % |

### Serious AE at Zinforo discontinuation

Yes

No

Unknown

### Seriousness criteria applied (for AEs indicated as serious)

Resulted in death

Life-threatening

Hospitalization/prolongation of hospitalization

Persistent/significant disability/incapacity

Congenital anomaly/birth defect

Important medical event

None of the above

Unknown

Abbreviations: AE: adverse event.

### Table 27. Post Zinforo treatment-Summary across all lines in patients with CAP

**Antibiotic treatment post Zinforo** 

All CAP patients (N=XX)

n %

#### Antibiotic treatment received for index infection after Zinforo

No

#### Post Zinforo treatment received

Aminoglycoside

Betalactam

Carbapenem

Ceftriaxone

Cephalosporins

Glycopeptide

Macrolide

Betalactam

/Combination

Quinolone

Sulfonamide

Clindamycin

Linezolid

Other antibiotic agent

Unknown

### Line of therapy

First

Second

Third

Fourth

### Number of post Zinforo lines of therapy

Mean (SD)

Median (Min-Max)

### Route of administration

Oral

Intra-venous

Intra-muscular

Subcutaneous

Unknown

### Duration from Zinforo discontinuation to initiation of new treatment (days)

Mean (SD)

Median (Min-Max)

Unknown

### **Duration of treatment (days)**


### Antibiotic treatment post Zinforo

All CAP patients (N=XX) n %

Mean (SD)

Median (Min-Max)

Unknown

### Treatment type

Empiric

Definitive/Specific

Unknown

### Number of administrations

Mean (SD)

Median (Min-Max)

### Number of doses administered

Mean (SD)

Median (Min-Max)

### **Administration location**

ICU

General ward

Unknown

### Reason for switch

Lack of efficacy of previous treatment

Side effect of previous treatment

Drug interaction of previous treatment

Results of susceptibility test/pathogen identification

Special population with renal impairment

Other

Unknown

Abbreviations: ICU: intensive care unit; Max: maximum; Min: minimum; SD: standard deviation.

### Table 28. Response to post-Zinforo treatment in patients with CAP

| Post Zinforo treatment response | All CAP patients (N=XX) |
|---------------------------------|-------------------------|
| | n % |

### Treatment response to post- Zinforo treatment

Clinical response

Clinical failure

Unknown

### Clinical cure achieved

Yes

No

Unknown

### If clinical failure to post-Zinforo treatment

Treatment modification due to adverse event

Drug-drug interaction

Insufficient response

Relapse/reoccurrence

Death due to infection

Death due to other

Unknown

#### **ANALYSES OF CSSTI PATIENTS** 8.1.8

### 8.1.9 PATIENT CHARACTERISTICS IN PATIENTS WITH CSSTI

Table 29. Demographic characteristics of included cSSTI patients at index hospitalization

```
Demographic characteristics
                                                                          All cSSTI patients (N=XX)
                                                                                 n
Age
  <90 years
  ≥ 90 years
  If <90 years,
     Mean (SD)
     Median (Min Max)
  <65 years
  ≥ 65 years
Sex
  Male
  Female
Race, Ethnicity
  White, Caucasian
  Black/African-American/Caribbean
  Latin-American
  Asian
  Middle Eastern
  Mixed
  Other
  Not available
Country
  France
  Greece
  Italy
  Spain
  Russia
  Brazil
  Columbia
  Mexico
Height (cm)
  Mean (SD)
  Median (Min-Max)
  Unknown
Weight (kg)
  Mean (SD)
  Median (Range)
  Unknown
BMI
  Mean (SD)
  Median (Min-Max)
```

Demographic characteristics

All cSSTI patients (N=XX)

n %

Unknown

Type of residence/cohabitation (pre index

if changed after discharge)

Nursing home or extended care facility

Living independently

Living with care support (family, friend, hired support)

Other

Unknown

**Smoking habits** 

Non-smoker

Ex-smoker (stopped ≥ 365 days ago)

Occasional smoker (less than 1 tobacco product per day)

Habitual smoker (1 or more tobacco products per day)

Unknown

Table 30. Medical history in patients with cSSTI

| Medical history | All cSSTI patients (N=XX) |
|-----------------|---------------------------|
| | n % |

# Medical condition(s) the patient presented at index visit hospitalization

None

AIDS/HIV infection

If HIV infected: Controlled with HAART

Yes (n, % HIV infected) No (n, % HIV infected) Unknown (n, % HIV infected)

Alcohol abuse

Cancer/malignancy

Cerebrovascular disease

Chronic dialysis within the past 30 days

Chronic obstructive pulmonary disease

Chronic renal disease

Congestive heart failure

Decompensated cirrhosis

Diabetes mellitus

Immunosuppressive disease

Influenza

Injection drug use

End stage liver disease

Peripheral vascular disease

Respiratory disease

Other relevant condition(s) or disease(s) requiring chronic drug

treatment.

Unknown

Abbreviations: AIDS/ HIV acquired immunodeficiency syndrome/ human immunodeficiency virus, HAART highly active antiretroviral therapy.

# Table 31. Hospitalization and treatments in the 3 months prior to index hospitalization in patients with cSSTI

| Prior hospitalization | All cSSTI patients (N=XX) |
|-----------------------|---------------------------|
| | n % |

Hospitalization for any reason in the 3 months before index hospitalization

Yes

No

Unknown

If hospitalized

Duration of Hospitalization previous to index

Mean (SD)

Median (Min-Max)

Invasive major surgical treatment in the 3 months before index

Yes

No

Unknown

Therapies received in the 3 months before index

Antimicrobial (e.g. antibiotics, antivirals)

Immunosuppressors/ immunomodulators

Anticoagulants

Non-steroid anti-inflammatory agents (NSAIs)

Home infusion therapy

Home wound care provided by a medical professional

Vone

### Table 32. cSSTI Characteristics

| Characteristics | All cSSTI patients | |
|-----------------|--------------------|---|
| | (N=XX) | |
| | n | % |

### Lesions involved in the patient's cSSTI

Abscess

Cellulitis/fasciitis

Post-traumatic wound

Post-surgical wound

Decubitus ulcer

Diabetic leg ulcer

Peripheral vascular disease ulcer

Burn

Bite

Unknown

None of the above

### Body areas involved in cSSTI

Head

Hand

Upper extremities

Lower extremities

Thorax

Abdomen

Genitalia

Unknown

Muscle

Unknown

### Extension of the skin infection (cm<sup>2</sup>)

<5 cm2

5-10 cm2

10-50 cm2

>50 cm2

Unknown

### Level of infection

Superficial

Deep incisional

Organ or space infection

Unknown

### **Anatomical structures affected**

Epithelium

Epidermis

Dermis

Subcutaneous fat


انانا

| Characteristics | All cSSTI patient<br>(N=XX) | S |
|-----------------|-----------------------------|---|
| | n | % |
| Fascia | | |
| Muscle | | |
| Unknown | | |

# Table 33. Diagnosis and infection details in patients with cSSTI

| Characteristics | All cSSTI patients |
|-----------------|--------------------|
| | (N=XX) |
| | n % |

### Time of cSSTI diagnosis

Prior to index hospitalization

Days prior to index hospitalization

Mean (SD)

Median (Min-Max)

During index hospitalization

Days prior after hospitalization (admission)

Mean (SD)

Median (Min-Max)

Unknown

### **Recurrent cSSTI infection**

Yes No Unknown

# **Table 34. cSSTI Diagnostics**

# Diagnostic criteria All cSSTI patients (N=XX) n %

### Triggering signs and symptoms for cSSTI at diagnosis

Purulent or seropurulent drainage/discharge

Bullae

Erythema

Fluctuance

Heat/localized warmth

Pain/tenderness to palpitation

Swelling/induration

Skin necrosis

### Systemic signs of cSSTI at diagnosis

Temperature > 38∘C

White blood cell count > 10,000/mm3 or < 4,500/mm3 or immature neutrophilis >10%

Septic shock

Organ dysfunction

Unknown

None of the above

### Tests conducted for cSSTI diagnosis

Blood cultures

Superficial swab and culture

Needle aspiration

Skin biopsy

Surgical sample

X-ray

Ultrasound

CT/MRI

Unknown/not performed

### Microbiological cSSTI diagnosis positive for

Methicillin resistance Staphylococcus aureus

Methicillin susceptible S. aureus (MSSA)

Staphylococcus coagulase negative

Vancomycin Intermediate S. aureus (VISA)

Streptococcus pneumonia

Multidrug resistant S. pneumoniae (MDRSP)

Penicillin resistant S. pneumoniae (PRSP)

Beta-hemolytic Streptococci

Streptococcus pyogenes

Streptococcus agalactiae

Enterococcus faecalis

Enterococcus faecium

Gram-negative bacilli

Non-fermenting enterobacteria


CCI

| Diagnostic criteria | All cSSTI patients (N=XX) |
|---------------------------------|---------------------------|
| | n % |
| Clostirdium spp. | |
| Other strict anaerobic bacteria | |
| Other microorganism | |
| Mixed flora | |
| Unknown | |
| None of the above | |

# 8.1.10 HEALTHCARE RESOURCE USE FOR CSSTI PATIENTS STARTING ZINFORO

### Table 35. Utilization during index hospitalization in patients with cSSTI

Resource utilization

All cSSTI patients (N=XX)

n %

### **Duration of index hospitalization** (days)

Mean (SD)

Median (Min-Max)

### **Duration of days in ICU**

Mean (SD)

Median (Min-Max)

### Quick sepsis-related organ failure assessment (qSOFA) conducted

Yes

No

Unknown

If qSOFA was conducted

(n, % of qSOFA assessed)

Glasgow coma scale <15

Systolic blood pressure <100 mmHg

High respiration rate (≥ 22 breaths per minute)

### Patient required isolation

Yes

No

Unknown

If patient isolated:

Duration of isolation (days)

Mean (SD)

Median (Min-Max)

Unknown

Abbreviations: ICU: intensive care unit; Max: maximum; Min: minimum; qSOFA: Quick sepsis-related organ failure assessment; SD: standard deviation.

### Table 36. Hospitalisation cost in patients with cSSTI

| Hospital Cost | All cSSTI patients (N=XX) |
|---------------|---------------------------|
| | n % |

### Hospital Cost - standard hospital (local currency)

Mean (SD)

Median (Min-Max)

### Hospital Cost - advanced level (local currency)

Mean (SD)

Median (Min-Max)

### Hospital Cost - standard hospital (USD)

Mean (SD)

Median (Min-Max)

### Hospital Cost - advanced level (USD)

Mean (SD)

Median (Min-Max)

Abbreviations: USD: US Dollars, Max: maximum; Min: minimum; SD: standard deviation.

Table 37. Utilization during index hospitalization by response status in patients with cSSTI

| Resource utilization | cSSTI respor<br>(N=XX) | iders | cSSTI no<br>responde<br>(N=XX) | ers |
|---|---|---|---|---|
| | n % | o I | n % | |

### **Duration of index hospitalization** (days)

Mean (SD)

Median (Min-Max)

### **Duration of days in ICU**

Mean (SD)

Median (Min-Max)

# Quick sepsis-related organ failure assessment (qSOFA) conducted

Yes

No

Unknown

If qSOFA was conducted

(n, % of qSOFA assessed)

Glasgow coma scale <15

Systolic blood pressure <100 mmHg

High respiration rate (≥ 22 breaths per

minute)

### Patient required isolation

Yes

No

Unknown

If patient isolated:

Duration of isolation (days)

Mean (SD)

Median (Min-Max)

Unknown

Table 38. Hospitalisation cost by response status in patients with cSSTI

| Hospital Cost | cSSTI responders<br>(N=XX) | cSSTI non-<br>responders<br>(N=XX) |
|---|---|---|
| | n % | n % |

### Hospital Cost- standard hospital (local currency)

Mean (SD)

Median (Min-Max)

### Hospital Cost- advanced level (local currency)

Mean (SD)

Median (Min-Max)

### Hospital Cost- standard hospital (USD)

Mean (SD)

Median (Min-Max)

### Hospital Cost- advanced level (USD)

Mean (SD)

Median (Min-Max)

Abbreviations: USD: US Dollars, Max: maximum; Min: minimum; SD: standard deviation.

### Table 39. Ventilation and parenteral nutrition in patients with cSSTI

Ventilation and parenteral nutrition

All cSSTI patients (N=XX)

n %

### Patient required mechanical ventilation

Yes

No

Unknown

If patient received ventilation:

### Type of ventilation

Invasive ventilation (n, % ventilated)

Duration of invasive ventilation (days)

Mean (SD)

Median (Min-Max)

Non-invasive ventilation (n, % ventilated)

Duration of non-invasive ventilation (days)

Mean (SD)

Median (Min-Max)

Including high flow oxygen therapy

Yes (n, % ventilated)

No (n, % ventilated)

Unknown (n, % ventilated)

### Patient received parenteral nutrition

Yes

No

Unknown

If Yes:

Duration of parenteral nutrition (days)

Mean (SD)

Median (Min-Max)

Unknown

Table 40. Treatments received during index hospitalization in patients with cSSTI

# Treatments received All cSSTI patients (N=XX) n %

### Treatment received during index hospitalization

Surgery related to the infection

Surgery unrelated to the infection

Blood pressure support

If blood pressure support received:

Fluid resuscitation (n,% blood pressure support)

Vasopressors (n,% blood pressure support)

Invasive procedures (n,% blood pressure support)

Unknown

Other

None of the above

### Table 41. Complications during index hospitalization in patients with cSSTI

Complications

All cSSTI patients (N=XX)

n %

### Renal failure necessitating renal replacement

Yes
No
Unknown
If renal replacement:
Duration of therapy (days)
Mean (SD)
Median (Min-Max)
Renal replacement after first dose of Zinforo
Yes (n,% with renal replacement)
No (n,% with renal replacement)
Unknown (n,% with renal replacement)
Serum creatinine at the first Zinforo dose (mg/dL)
Mean (SD)
Median (Min-Max)

### Complications developed during index hospitalization

Sepsis Severe sepsis Septic shock Unknown None of the above

Unknown

# Table 42. Dosages of Zinforo and other antibiotics in patients with cSSTI

Complications

All cSSTI patients (N=XX)

n %

### Total number of doses of Zinforo administered

Mean (SD) Median (Min-Max)

# Total number doses of other antibiotics administered in combination with Zinforo

Mean (SD) Median (Min-Max)

# Total number of doses of other antibiotics administered post Zinforo treatment

Mean (SD) Median (Min-Max)

### Table 43. Resource use post index hospitalization in patients with cSSTI

```
Resource utilization post index hospitalization
                                                                             All cSSTI patients (N=XX)
                                                                                        n %
Home-based care received through a health-care agency (e.g. for
wounds, intravenous infusions)
  Yes
  No
  Unknown
  If home based care received,
     Duration of home-based care (days)
         Mean (SD)
         Median (Min-Max)
Re-hospitalized within 30 days of initial discharge
  Yes
  No
  Unknown
  If re-hospitalized,
     Number of re-hospitalizations
         Mean (SD)
         Median (Min-Max)
     Duration of all hospitalizations
         Mean (SD)
         Median (Min-Max)
     Admission reason:
         For index infection (n,% of re-hospitalizations)
         For other reason (n,% of re-hospitalizations)
```

Abbreviations: Max: maximum; Min: minimum; SD: standard deviation.

Unknown (n,% of re-hospitalizations)

# 8.1.11 PHYSICIANS USE OF ZINFORO® (AND OTHER ANTIBIOTICS) DURING INDEX HOPSPITALIZATION IN PATIENTS WITH CSSTI

# Table 44. Pre Zinforo treatment- Summary across all treatment lines in patients with cSSTI

| Antibiotic treatment pre Zinforo | All cSSTI patients (N=XX) |
|----------------------------------|---------------------------|
| Antibiotic treatment pre Zimoro | All Coott patients (N-AA) |
| | n % |

### Antibiotic treatment for the index infection received prior to

Zinforo

Yes

No

#### Pre Zinforo treatment received

Aminoglycoside

Betalactam

Carbapenem

Ceftriaxone

Cephalosporins

Glycopeptide

Macrolide

Betalactam

/Combination

Quinolone

Sulfonamide

Clindamycin

Linezolid

Other antibiotic agent

Unknown

### Line of therapy

First

Second

Third

Fourth

### Number of pre Zinforo lines of therapy

Mean (SD)

Median (Min-Max)

### Route of administration

Oral

Intra-venous

Intra-muscular

Subcutaneous

Unknown


انانا

### **Antibiotic treatment pre Zinforo**

All cSSTI patients (N=XX) n %

### **Duration of pre Zinforo treatment (days)**

Mean (SD)

Median (Min-Max)

### Treatment type

Empiric

Definitive/Specific

Unknown

### Number of administrations

Mean (SD)

Median (Min-Max)

### Number of doses administered

Mean (SD)

Median (Min-Max)

#### **Administration location**

ICU

General ward

At home

Out patient

Medical setting

Unknown

### **Treatment modification**

Yes

No

Unknown

If yes:

Time to treatment modification from initial dose

Reason for treatment modification

Treatment response

Time to clinical response

Clinical failure details

Daily dose unit

Table 45. Pre Zinforo treatment by line of treatment in patients with cSSTI

| Pre Zinforo treatment | | Line of treatment | | |
|------------------------|----------|-------------------|----------|----------|
| | 1st Line | 2nd Line | 3rd Line | 4th Line |
| | N, % | N, % | N, % | N, % |
| Aminoglycoside | | | | |
| Betalactam | | | | |
| Carbapenem | | | | |
| Ceftriaxone | | | | |
| Cephalosporins | | | | |
| Glycopeptide | | | | |
| Macrolide | | | | |
| Betalactam | | | | |
| /Combination | | | | |
| Quinolone | | | | |
| Sulfonamide | | | | |
| Clindamycin | | | | |
| Linezolid | | | | |
| Other antibiotic agent | | | | |
| Unknown | | | | |

### Table 46. Zinforo treatment during index hospitalization in patients with cSSTI

Zinforo treatment

All cSSTI patients (N=XX)

n %

### Zinforo line of therapy

First

Second

Third

Fourth

### **Duration of Zinforo treatment (days)**

Mean (SD)

Median (Min-Max)

Unknown

### Time from admission to 1st dose (days)

Mean (SD)

Median (Min-Max)

Unknown

### Time from symptom onset to 1st dose (days)

Mean (SD)

Median (Min-Max)

Unknown

### Treatment type

Empiric

Definitive/Specific

Unknown

### Daily dose (mg/kg)

Mean (SD)

Median (Min-Max)

### Number of infusions per day

Mean (SD)

Median (Min-Max)

Unknown

#### Administration location

ICU

General ward

At home

Out-patient setting

Medical clinic

Unknown

Abbreviations: ICU: intensive care unit; Max: maximum; Min: minimum; SD: standard deviation.


CCI

### Table 47. Zinforo administered in combination therapy in patients with cSSTI

Antibiotic treatments given in combination with Zinforo

All cSSTI patients (N=XX)

n %

#### Zinforo as Mono/ Combination treatment

Monotherapy Combination therapy Unknown

#### If administered in combination:

#### Antibiotic treatment received

Aminoglycoside

Betalactam

Carbapenem

Ceftriaxone

Cephalosporins

Glycopeptide

Macrolide

Betalactam

/Combination

Quinolone

Sulfonamide

Clindamycin

Linezolid

Other antibiotic agent

Unknown

### Route of administration

Oral

Intra-venous

Intra-muscular

Subcutaneous

Unknown

### **Duration of combination treatment (days)**

Mean (SD)

Median (Min-Max)

Unknown

### Number of doses administered

Mean (SD)

Median (Min-Max)

Unknown

Abbreviations: Max: maximum; Min: minimum; SD: standard deviation.

# Table 48. Zinforo treatment and concomitant therapy in patients with cSSTI

| | 1 3 1 |
|-------------------------------------|---------------------------|
| Therapies concomitant to Zinforo | All cSSTI patients (N=XX) |
| | n % |
| Concomitant therapy given | |
| Yes | |
| No | |
| If concomitant therapy "yes" | |
| Therapy received | |
| Immunosuppressors/ Immunomodulators | |

Anticoagulants
Non-steroidal anti-inflammatory agents (NSAIs)

Chemotherapeutic agents

Other Unknown

## 8.1.12 TREATMENT RESPONSE TO ZINFORO® IN PATIENTS WITH CSSTI

# Table 49. Response to Zinforo treatment in patients with cSSTI

All cSSTI patients (N=XX) Treatment response n %

# Zinforo treatment response

Clinical response Clinical failure Time to clinical response Mean (SD)

Median (Min-Max)

Unknown

## Zinforo early treatment response

Response ≤3 days Response >3days No response Unknown

#### Clinical cure achieved

Yes No

Time to clinical cure

Mean (SD)

Median (Min-Max)

Unknown

## Reduction of ≥20% from baseline area achieved

Time to ≥20% reduction from baseline area

Mean (SD)

Median (Min-Max)

Unknown

# Cessation of spread measured by total infection area

Time to cessation of spread

Mean (SD)

Median (Min-Max)

Unknown

# Cessation of spread measured by infection length and width

Time to cessation of spread

Mean (SD)

Median (Min-Max)

Unknown

Abbreviations: Max: maximum; Min: minimum; SD: standard deviation.


## 8.1.13 ADDITIONAL CLINICAL OUTCOMES IN PATIENTS WITH CSSTI

# Table 50. Additional clinical outcomes in response to Zinforo treatment in patients with cSSTI

# Additional clinical outcomes All cSSTI patients (N=XX) n %

## Discharge status

Died in the hospital

Discharged to a nursing home or extended care facility

Discharged to independent living (with or without support)

Other

Unknown

#### Vital status at end of follow up

Patient is still alive

Patient is deceased

If deceased

Duration of days from discharge until death(days)

Mean (SD)

Median (Min-Max)

Unknown

# Minimum inhibitory concentrations (MIC) of antibacterial drugs assessed

Yes

No

Unknown

If assessed

Day of assessment since index hospitalization

Mean (SD)

Median (Min-Max)

MIC of ceftaroline for all isolated pathogens

MIC of oxacillin, vancomycin, linezolid, and daptomycin for S. aureus

MIC of ceftriaxone for MSSA

MIC of penicillin and ceftriaxone for S. pneumonia

Abbreviations: Max: maximum; MIC: minimum inhibitory concentrations; Min: minimum; SD: standard deviation.

# 8.1.14 TREATMENT MODIFICATIONS / ADVERSE EVENTS IN PATIENTS WITH CSSTI

# Table 51. Clinical failure with Zinforo in patients with cSSTI

| Clinical failure with Zinforo | All cSSTI patients (N=XX) |
|-------------------------------|---------------------------|
| | n % |

# Etiology of clinical failure

Failure related to cSSTI Failure unrelated to cSSTI Unknown

#### Reason for clinical failure

Treatment modification due to AE Time to modification (days)

Mean (SD)

Median (Min-Max)

Unknown

Drug-drug interaction

Insufficient response

Death due to index infection

Time to death due to infection (days)

Mean (SD)

Median (Min-Max)

Death due to other

Relapse or recurrence

Time to relapse/recurrence:

Mean (SD)

Median (Min-Max)

Unknown

Abbreviations: AE: adverse events; Max: maximum; Min: minimum; SD: standard deviation.

# Table 52. Clinical failure with Zinforo due to adverse events in patients with cSSTI

Clinical failure to Zinforo due to AEs

All cSSTI patients (N=XX)

n %

## AE causing Zinforo discontinuation

Infections and infestations

Clostridium difficile colitis

Other

Blood and lymphatic system disorders

Activated partial thromboplastin time (aPTT) prolonged

Agranulocytosis

Anaemia

Eosinophilia

International normalized ratio (INR) increased

Leucopenia

Neutropenia

Prothrombin time (PT) prolonged

Thrombocytopenia

Other

Immune system disorders

Anaphylaxis

Hypersensitivity (e.g. urticarial, lip and face swelling)

Pruritus

Rash

Other

Nervous system disorders

Dizziness

Headache

Other

Vascular disorders

Phlebitis

Other

Gastrointestinal disorders

Abdominal pain

Diarrhea

Nausea

Vomiting

Other

Hepatobiliary disorders

Increased transaminases

Other

Renal urinary disorders

Blood creatinine increased

Other

General disorders and administrative site conditions

Infusion site reaction (e.g. erythema, phlebitis, pain)

Pyrexia

Other

Investigations


CCI

# Clinical failure to Zinforo due to AEs Coombs direct test positive All cSSTI patients (N=XX) n %

Other Unknown

Abbreviations: AE: adverse events, aPTT: activated partial thromboplastin time

# Table 53. Seriousness of adverse events in patients with cSSTI

| Clinical failure to Zinfore | All cSSTI patients (N=XX) |
|-----------------------------|----------------------------|
| Clinical failure to Zinforo | All C5511 batterits (N-AA) |
| | , |
| | n % |
| | II /0 |

# Serious AE at Zinforo discontinuation

Yes

No

Unknown

# Seriousness criteria applied (for AEs indicated as serious)

Resulted in death

Life-threatening

Hospitalization/prolongation of hospitalization

Persistent/significant disability/incapacity

Congenital anomaly/birth defect

Important medical event

None of the above

Unknown

Abbreviations: AE: adverse event.

# Table 54. Post Zinforo treatment- Summary across all lines in patients with cSSTI

Antibiotic treatment post Zinforo

All cSSTI patients (N=XX)

n %

#### Antibiotic treatment received for index infection after Zinforo

Yes

No

#### Post Zinforo treatment received

Aminoglycoside

Betalactam

Carbapenem

Ceftriaxone

Cephalosporins

Glycopeptide

Macrolide

Betalactam

/Combination

Quinolone

Sulfonamide

Clindamycin

Linezolid

Other antibiotic agent

Unknown

# Line of therapy

First

Second

Third

Fourth

# Number of post Zinforo lines of therapy

Mean (SD)

Median (Min-Max)

## Route of administration

Oral

Intra-venous

Intra-muscular

Subcutaneous

Unknown

# Duration from Zinforo discontinuation to initiation of new treatment (days)

Mean (SD)

Median (Min-Max)

Unknown

# **Duration of treatment (days)**


CCI

# Antibiotic treatment post Zinforo

All cSSTI patients (N=XX) n %

Mean (SD)

Median (Min-Max)

Unknown

## Treatment type

Empiric

Definitive/Specific

Unknown

## Number of administrations

Mean (SD)

Median (Min-Max)

# Number of doses administered

Mean (SD)

Median (Min-Max)

#### **Administration location**

ICU

General ward

Unknown

## Reason for switch

Lack of efficacy of previous treatment

Side effect of previous treatment

Drug interaction of previous treatment

Results of susceptibility test/pathogen identification

Special population with renal impairment

Other

Unknown

Abbreviations: ICU: intensive care unit; Max: maximum; Min: minimum; SD: standard deviation.

# Table 55. Response to post-Zinforo treatment in patients with cSSTI

| Post Zinforo treatment response | All cSSTI patients (N=XX) |
|---------------------------------|---------------------------|
| | n % |

# Treatment response to post- Zinforo treatment

Clinical response

Clinical failure

Unknown

## Clinical cure achieved

Yes

No

Unknown

# If clinical failure to post-Zinforo treatment

Treatment modification due to adverse event

Drug-drug interaction

Insufficient response

Relapse/reoccurrence

Death due to infection

Death due to other

Unknown

## 9 REFERENCES

- 1. Martinez R, Reyes S, Lorenzo MJ, Menendez R. Impact of guidelines on outcome: the evidence. *Semin Respir Crit Care Med.* 2009;30(2):172-178.
- 2. Welte T. Managing CAP patients at risk of clinical failure. *Respir Med.* 2015;109(2):157-169.
- 3. Personne V, Chevalier J, Buffel du Vaure C, Partouche H, Gilberg S, de Pouvourville G. CAPECO: Cost evaluation of community acquired pneumonia managed in primary care. *Vaccine*. 2016;34(19):2275-2280.
- 4. Rozenbaum MH, Mangen MJ, Huijts SM, van der Werf TS, Postma MJ. Incidence, direct costs and duration of hospitalization of patients hospitalized with community acquired pneumonia: A nationwide retrospective claims database analysis. *Vaccine*. 2015;33(28):3193-3199.
- 5. Kolditz M, Tesch F, Mocke L, Hoffken G, Ewig S, Schmitt J. Burden and risk factors of ambulatory or hospitalized CAP: A population based cohort study. *Respir Med.* 2016;121:32-38.
- 6. Schnoor M, Hedicke J, Dalhoff K, Raspe H, Schafer T, group Cs. Approaches to estimate the population-based incidence of community acquired pneumonia. *J Infect*. 2007;55(3):233-239.
- 7. Ramirez JA, Anzueto AR. Changing needs of community-acquired pneumonia. *J Antimicrob Chemother.* 2011;66 Suppl 3:iii3-9.
- 8. Blasi F, Garau J, Medina J, et al. Current management of patients hospitalized with community-acquired pneumonia across Europe: outcomes from REACH. *Respir Res.* 2013;14:44.
- 9. Capelastegui A, Espana PP, Bilbao A, et al. Etiology of community-acquired pneumonia in a population-based study: link between etiology and patients characteristics, process-of-care, clinical evolution and outcomes. *BMC Infect Dis.* 2012:12:134.
- 10. Dryden MS. Complicated skin and soft tissue infection. *J Antimicrob Chemother*. 2010;65 Suppl 3:iii35-44.
- 11. Raghavan M, Linden PK. Newer treatment options for skin and soft tissue infections. *Drugs*. 2004;64(15):1621-1642.
- 12. Tognetti L, Martinelli C, Berti S, et al. Bacterial skin and soft tissue infections: review of the epidemiology, microbiology, aetiopathogenesis and treatment: a collaboration between dermatologists and infectivologists. *J Eur Acad Dermatol Venereol.* 2012;26(8):931-941.
- 13. Hatoum HT, Akhras KS, Lin SJ. The attributable clinical and economic burden of skin and skin structure infections in hospitalized patients: a matched cohort study. *Diagn Microbiol Infect Dis.* 2009;64(3):305-310.

- 14. Talan DA, Salhi BA, Moran GJ, et al. Factors associated with decision to hospitalize emergency department patients with skin and soft tissue infection. *West J Emerg Med.* 2015;16(1):89-97.
- 15. Lodise TP, Fan W, Sulham KA. Hospital admission patterns in adult patients with skin and soft tissue infections: Identification of potentially avoidable hospital admissions through a retrospective database analysis. *Hosp Pract (1995)*. 2015;43(3):137-143.
- 16. Garau J, Ostermann H, Medina J, et al. Current management of patients hospitalized with complicated skin and soft tissue infections across Europe (2010-2011): assessment of clinical practice patterns and real-life effectiveness of antibiotics from the REACH study. *Clin Microbiol Infect*. 2013;19(9):E377-385.
- 17. Lipsky BA, Weigelt JA, Gupta V, Killian A, Peng MM. Skin, soft tissue, bone, and joint infections in hospitalized patients: epidemiology and microbiological, clinical, and economic outcomes. *Infect Control Hosp Epidemiol*. 2007;28(11):1290-1298.
- 18. File TM, Jr., Low DE, Eckburg PB, et al. FOCUS 1: a randomized, double-blinded, multicentre, Phase III trial of the efficacy and safety of ceftaroline fosamil versus ceftriaxone in community-acquired pneumonia. *J Antimicrob Chemother*. 2011;66 Suppl 3:iii19-32.
- 19. Low DE, File TM, Jr., Eckburg PB, et al. FOCUS 2: a randomized, double-blinded, multicentre, Phase III trial of the efficacy and safety of ceftaroline fosamil versus ceftriaxone in community-acquired pneumonia. *J Antimicrob Chemother*. 2011;66 Suppl 3:iii33-44.
- 20. Ramani A, Udeani G, Evans J, et al. Contemporary use of ceftaroline fosamil for the treatment of community-acquired bacterial pneumonia: CAPTURE study experience. *Journal of chemotherapy (Florence, Italy)*. 2014;26(4):229-234.
- 21. Eckberg PF, D. Llorens, L. Smith, A. Witherell, G. Laudano, J. Thye, D. Day 4 clinical response of ceftaroline for community-acquired bacterial pneumonia. *Infectious Diseases in Clinical Practice*. 2012;20(4):254-260.
- 22. File TM, Jr., Wilcox MH, Stein GE. Summary of ceftaroline fosamil clinical trial studies and clinical safety. *Clin Infect Dis.* 2012;55 Suppl 3:S173-180.
- 23. Wilcox MH, Corey GR, Talbot GH, et al. CANVAS 2: the second Phase III, randomized, double-blind study evaluating ceftaroline fosamil for the treatment of patients with complicated skin and skin structure infections. *J Antimicrob Chemother*. 2010;65 Suppl 4:iv53-iv65.
- 24. Corey GR, Wilcox MH, Talbot GH, et al. CANVAS 1: the first Phase III, randomized, double-blind study evaluating ceftaroline fosamil for the treatment of patients with complicated skin and skin structure infections. *J Antimicrob Chemother*. 2010;65 Suppl 4:iv41-51.
- 25. Corey GR, Wilcox M, Talbot GH, et al. Integrated analysis of CANVAS 1 and 2: phase 3, multicenter, randomized, double-blind studies to evaluate the safety and efficacy of ceftaroline versus vancomycin plus aztreonam in complicated skin and skin-structure infection. *Clin Infect Dis.* 2010;51(6):641-650.

26. Dryden M, Zhang Y, Wilson D, Iaconis JP, Gonzalez J. A Phase III, randomized, controlled, non-inferiority trial of ceftaroline fosamil 600 mg every 8 h versus vancomycin plus aztreonam in patients with complicated skin and soft tissue infection with systemic inflammatory response or underlying comorbidities. *J Antimicrob Chemother*. 2016;71(12):3575-3584.